CLINICAL TRIAL: NCT03544684
Title: Fasted High-Intensity Interval and Moderate-Intensity Continuous Exercise Are Not Associated With A Detrimental 24-Hour Blood Glucose Profile
Brief Title: Fasted Exercise in People With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Sam Shepherd, Lecturer/Senior Lecturer, Principle Investigator, Liverpool John Moores University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: T1D_PARTA
Record Dates: First submitted 2018-05-09; First posted 2018-06-04 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control day with no exercise (Experimental): glycaemic profile will be assessed using continuous glucose monitors following a single 24-hour period in which participants performed no exercise
  Interventions: Behavioral: Effects of the type of exercise on blood glucose concentrations
- High intensity interval training (HIT) (Experimental): glycaemic profile will be assessed using continuous glucose monitors following a 24-hour period whereby participants performed a single bout of high-intensity interval training (HIT) in the morning under fasted conditions
  Interventions: Behavioral: Effects of the type of exercise on blood glucose concentrations
- moderate intensity continuous training (MICT) (Experimental): glycaemic profile will be assessed using continuous glucose monitors following a 24-hour period whereby participants performed a single bout of moderate-intensity continuous training (MICT) in the morning under fasted conditions
  Interventions: Behavioral: Effects of the type of exercise on blood glucose concentrations

INTERVENTIONS:
Behavioral: Effects of the type of exercise on blood glucose concentrations — glucose concentrations were assessed over the 24 hour periods following no exercise, a single bout of high intensity interval training and a single bout of moderate intensity continuous training

SUMMARY:
This study aims to compare the effect of a bout of high-intensity interval training (HIT) with a bout of moderate-intensity continuous training (MICT) on glucose concentrations over the subsequent 24h period.

DETAILED DESCRIPTION:
This study aims to compare the effect of a bout of high-intensity interval training (HIT) with a bout of moderate-intensity continuous training (MICT) on glucose concentrations over the subsequent 24h period. Fourteen people with type 1 diabetes (duration of type 1 diabetes 8.2±1.4 years), all on basal-bolus regimen, completed a randomised, counterbalanced, crossover study. Continuous glucose monitoring was used to assess glycaemic control following a single bout of HIT (6 x 1min intervals) and 30 mins of moderate-intensity continuous training (MICT) on separate days, compared to a non-exercise control day (CON). Exercise was undertaken following an overnight fast with omission of short-acting insulin. Capillary blood glucose samples were recorded pre and post-exercise to assess the acute changes in glycaemia during HIT and MICT.

ELIGIBILITY:
Inclusion Criteria:

* duration of type 1 diabetes >6 months
* basal bolus regimen
* no significant history of hyper- or hypoglycaemia (determined from medical history

Exclusion Criteria:

* duration of type 1 diabetes <6 months,
* insulin pump therapy
* significant history of hyper- or hypoglycaemia (determined from medical history)
* obesity (BMI >30 kg∙m-2)
* pregnancy or planning pregnancy, uncontrolled hypertension (>180/100 mmHg)
* angina
* autonomic neuropathy
* taking any medication that affects heart rate
* major surgery planned within 6 weeks of the study
* severe nonproliferative and
* unstable proliferative retinopathy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
24 hour glycaemic profile | 24 hours
  Continuous glucose monitoring will be used to assess the effects of an acute bout of fasted high intensity interval training or moderate intensity continuous training on 24 hour glycaemic profile.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool John Moores University, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available to others

REFERENCES:
- [Derived] Scott SN, Cocks M, Andrews RC, Narendran P, Purewal TS, Cuthbertson DJ, Wagenmakers AJM, Shepherd SO. High-Intensity Interval Training Improves Aerobic Capacity Without a Detrimental Decline in Blood Glucose in People With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Feb 1;104(2):604-612. doi: 10.1210/jc.2018-01309. PMID 30281094
- [Derived] Scott SN, Cocks M, Andrews RC, Narendran P, Purewal TS, Cuthbertson DJ, Wagenmakers AJM, Shepherd SO. Fasted High-Intensity Interval and Moderate-Intensity Exercise Do Not Lead to Detrimental 24-Hour Blood Glucose Profiles. J Clin Endocrinol Metab. 2019 Jan 1;104(1):111-117. doi: 10.1210/jc.2018-01308. PMID 30252054